CLINICAL TRIAL: NCT03173339
Title: Influence of Remifentanil on Postoperative Sore Throat in Patients Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HighRemiSoreThroat
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-05

CONDITIONS: Hip Arthroplasty
Keywords: intubation; pharyngitis; remifentanil
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low remifentanil and high sevoflurane (Active Comparator): Remifentanil was administered as 0.1 mcg/kg/min. Sevoflurane was started as 0.5 MAC. Sevoflurane dose was adjusted to maintain blood pressure (20% of preoperative blood pressure) and bispectral index (40-60) by 0.2 %.
  Interventions: Procedure: Endotracheal intubation using laryngoscope; Drug: Low remifentanil; Drug: High sevoflurane
- High remifentanil and low sevoflurane (Experimental): Sevoflurane was administered as 0.5 MAC. Remifentanil was started as 0.25 mcg/kg/min. Remifentanil dose was adjusted to maintain blood pressure (20% of preoperative blood pressure) and bispectral index (40-60) by 0.05 mcg/kg/min.
  Interventions: Procedure: Endotracheal intubation using laryngoscope; Drug: High remifentanil; Drug: Low sevoflurane

INTERVENTIONS:
Procedure: Endotracheal intubation using laryngoscope — Endotracheal intubation was done using laryngoscope for general anesthesia.
Drug: High remifentanil — Remifentanil was started as 0.25 mcg/kg/min. Remifentanil dose was adjusted to maintain blood pressure (20% of preoperative blood pressure) and bispectral index (40-60) by 0.05 mcg/kg/min.
  Arms: High remifentanil and low sevoflurane
Drug: Low remifentanil — Remifentanil was administered as 0.1 mcg/kg/min.
  Arms: Low remifentanil and high sevoflurane
Drug: High sevoflurane — Sevoflurane was started as 0.5 MAC. Sevoflurane dose was adjusted to maintain blood pressure (20% of preoperative blood pressure) and bispectral index (40-60) by 0.2 %.
  Arms: Low remifentanil and high sevoflurane
Drug: Low sevoflurane — Sevoflurane was administered as 0.5 MAC.
  Arms: High remifentanil and low sevoflurane

SUMMARY:
This investigation is planned to compare the incidence and severity of postoperative sore throat according to the dose of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for general anesthesia with endotracheal intubation

Exclusion Criteria:

* Difficult airway
* Rapid sequence induction
* Recent sore throat
* Recent upper respiratory infection
* Asthma
* Chronic obstructive pulmonary disease
* Chronic cough
* Pregnancy
* Allergy to remifentanil
* Friable teeth
* History of head and neck surgery
* Multiple intubation attempts
* Regional anesthetic agents
* Gastric tube
* Dexamethasone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with sore throat | At 24 hr

SECONDARY OUTCOMES:
Number of participants with sore throat | At 0, 2, 4 and 24 hr
Number of participants with hoarseness | At 0, 2, 4 and 24 hr
Number of participants with cough | At 0, 2, 4 and 24 hr
Number of participants with nausea | At 0, 2, 4 and 24 hr
Number of participants with vomiting | At 0, 2, 4 and 24 hr
Number of participants with additional pain medication | At 0, 2, 4 and 24 hr
Visual analogue scale of postoperative pain | At 0, 2, 4 and 24 hr
Number of participants with shivering | At 0, 2, 4 and 24 hr
Requirements of analgesics | At 0, 2, 4 and 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Chang Kim, MD. Ph. D., Principal Investigator — Keimyung University
Locations (1):
- Keimyung University, Daegu, Non-US/Canada, South Korea

REFERENCES:
- [Derived] Park JH, Lee YC, Lee J, Kim H, Kim HC. The influence of high-dose intraoperative remifentanil on postoperative sore throat: a prospective randomized study: A CONSORT compliant article. Medicine (Baltimore). 2018 Dec;97(50):e13510. doi: 10.1097/MD.0000000000013510. PMID 30558006